CLINICAL TRIAL: NCT05680285
Title: Clinical and Radiographic Evaluation of Low Level Laser Therapy in Primary Tooth Pulpotomy Treatment
Brief Title: Evaluation of Low Level Laser Therapy in Primary Tooth Pulpotomy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UsakU10
Record Dates: First submitted 2022-12-16; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Pulpotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diode laser pulpotomy (Experimental): * Diode laser (Solase-976 Dental Diode Laser)
  * With a wavelength of 980 nm and a frequency of 110 Hz
  * In pulse mode, working for 1 ms and stopping for 8 ms
  * With a power output of 1 W during each laser pulse from the 400 µm fiber optic tip
  * By touching the fiber optic tip to the remaining pulp tissue
  * for 3 seconds
  * With 3 J energy to each root pulp during the process
  Interventions: Device: diode lazer
- low level diode laser pulpotomy (Experimental): * Diode laser (Solase-976 Dental Diode Laser)
  * It has a wavelength of 980 nm and a frequency of 165 Hz.
  * In pulse mode by setting it to run for 2 ms and stop for 4 ms
  * At a power of 0.2 W during each laser pulse from a 400 µm fiber optic tip
  * Without the fiber optic tip touching the remaining pulp tissue
  * for 10 seconds
  * With 2 J Energy to each root pulp
  Interventions: Device: low level diode laser

INTERVENTIONS:
Device: diode lazer — diode laser was applied during the pulpotomy procedure
  Arms: diode laser pulpotomy
Device: low level diode laser — Low-dose diode laser was applied during the pulpotomy procedure
  Arms: low level diode laser pulpotomy

SUMMARY:
In our study, it was aimed to compare the long-term effectiveness of diode laser and low level laser therapy and primary tooth amputation treatments using calcium hydroxide (LLLT+CH) in primary second molars with deep dentinal caries. Ninety patients ( 42 Gırl, 48 Boy) aged 6-9 years with deep dentin caries in the mandibular second molar were included in the study. The patients were randomly selected according to the treatment to be applied and divided into two groups as the diode laser group (N=45) and the LLLT+CH group (N=45). The patients were called for control appointments at the 1st, 3rd, 6th and 12th months after the treatment, and both clinical and radiographic follow-ups were performed. Chi-square and Fisher's Exact tests were used to compare categorical variables according to groups in statistical analysis, and p<0.05 was considered significant. When the study results at the end of 12 months were evaluated, the diode laser group had a clinical success rate of 95.6%, and a success rate of 93.3% radiologically; The LLLT+CH group had a success rate of 97.7% clinically and 90.9% radiologically. There was no statistically significant difference between the success rates of the groups (p>0.05). According to the clinical and radiographic results of our study, it was determined that diode laser and LLLT+CH amputations showed similar success rates in primary second molars with deep dentin caries. It has been seen that both methods can be used safely in primary tooth amputations. It is thought that clinical and histological studies and studies examining the effectiveness of dental laser applications in primary tooth amputation treatment are needed.

ELIGIBILITY:
Inclusion Criteria:

Clinical Criteria

* No systemic disease
* Not allergic to the materials used
* Children with scores of 1 and 2 according to the Frankel behavioral scale
* Those who have erupted permanent first molars
* The one in occlusion with the opposing tooth
* Not having bad oral habits
* No structural anomaly in the teeth
* No spontaneous or nocturnal pain
* No sensitivity to palpation or percussion
* Abscess and fistula formation free
* No pathological mobility
* During treatment, pulp bleeding is controlled within 5 minutes.
* With a crown that can be made of stainless steel crown (PÇK)

Radiographic Criteria

* Having a deep dentin caries lesion very close to the pulp
* No resorption in the bifurcation and periapical area
* Periodontal space is healthy and there is no periapical region pathology
* Absence of internal and external root resorption in roots
* No calcified masses in the pulp
* Teeth that did not exceed one-third of the physiological root resorption were included in the study.

Exclusion Criteria

-Children with a score of 1 and 4 on the Frankel Scale were excluded.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
radiographic success of treatments at the end of 12 months | 12 months
  teeth without any signs of pathological internal and external root resorption, enlargement of the periodontal space, and radiolucency in the periapical and furcation region
clinical success of treatments at the end of 12 months | 12 months
  teeth without any of the signs of spontaneous pain, tenderness on palpation and percussion, pathological mobility, sinus tract or gingival abscess form, lymphodanepathy in the relevant region

CONTACTS AND LOCATIONS:
Overall Officials: Tugba YIGIT, Principal Investigator — Uşak University
Locations (1):
- Usak University, Uşak, Turkey (Türkiye)